CLINICAL TRIAL: NCT03035383
Title: Purse String Suture for the Closure of Large Thyroidectomy Resulted in Better Cosmetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Kurnia, Head of Surgical Oncology, Dr Cipto Mangunkusumo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCiptoMGHAKurnia
Record Dates: First submitted 2017-01-22; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Thyroidectomy
Keywords: Large thyroid; purse string suture; thyroidectomy

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled study
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purse String Technique (Experimental): Thyroidectomy closure is performed using purse string technique.
  Interventions: Procedure: Purse string technique
- Conventional technique (Active Comparator): Thyroidectomy closure is performed using conventional technique.
  Interventions: Procedure: Conventional technique

INTERVENTIONS:
Procedure: Purse string technique — Thyroidectomy closure is performed using purse string suturing technique.
  Other Names: PST
  Arms: Purse String Technique
Procedure: Conventional technique — Thyroidectomy closure is performed using conventional suturing technique.
  Other Names: CT
  Arms: Conventional technique

SUMMARY:
Thyroidectomy for large thyroid tumor poses a problem of cosmetics, especially in terms of wide post-operative scar and prominent neck wrinkles. In this manuscript, we performed purse-string suture for the first time for the closure of skin defect after thyroidectomy of large thyroid tumors which resulted in better cosmetics as compared to the conventional suturing method.

DETAILED DESCRIPTION:
Increasing demand for better cosmetics following thyroidectomy for large thyroid tumor of > 6 cm diameter created a necessity to find an alternative to the conventional technique (CT), which could be addressed by purse string technique (PST). A non-randomized controlled trial was conducted to new thyroid tumor patients at Cipto Mangunkusumo Hospital (RSCM) from October 2013 until December 2014. Thirty patients grouped into two intervention arms of thyroidectomy with PST and CT were assessed for post-operative scar outcomes.

ELIGIBILITY:
Inclusion Criteria:

* New cases of thyroid tumor in Doctor Cipto Mangunkusumo General Hospital
* Tumor diameter > 6 cm

Exclusion Criteria:

* Previous surgery in the anterior neck area
* Local involvement of lymph nodes requiring nodes dissection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Length of scar | 8 to 12 weeks following thyroidectomy
  Length of scar in milimeter
Width of scar | 8 to 12 weeks following thyroidectomy
  Width of scar in milimeter
Wrinkle | 8 to 12 weeks following thyroidectomy
  Presence of wrinkle
Patient's satisfaction | 8 to 12 weeks following thyroidectomy
  Patient's satisfaction assessed using Likert scale of 1 to 10

SECONDARY OUTCOMES:
Duration of surgery | During surgery
  Duration of surgery in minutes
Bleeding | During surgery
  Volume of bleeding during surgery in cc
Post operative hospital stay | 1 week following thyroidectomy
  Post operative hospital stay

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.